CLINICAL TRIAL: NCT06876623
Title: A Single-dose, Two-sequence, Four-Period, Fully Replicated Crossover Bioequivalence Study of Dabigatran Etexilate Mesylate Capsules in Healthy Subjects Under Fasting and Fed Conditions
Brief Title: Bioequivalence Study of Two Dabigatran Etexilate Mesylate Capsules in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital Of Guizhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: YG-18007-BE
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-03

CONDITIONS: Bioequivalence of Dabigatran Etexilate Mesylate Capsules From Two Different Manufacturers in Healthy Chinese Subjects
MeSH Terms: interventions — Dabigatran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fasting TRTR group (Experimental)
  Interventions: Drug: dabigatran etexilate mesylate capsules 150mg
- Fasting RTRT group (Experimental)
  Interventions: Drug: dabigatran etexilate mesylate capsules 150mg
- Postprandial TRTR group (Experimental)
  Interventions: Drug: dabigatran etexilate mesylate capsules 150mg
- Postprandial RTRT group (Experimental)
  Interventions: Drug: dabigatran etexilate mesylate capsules 150mg

INTERVENTIONS:
Drug: dabigatran etexilate mesylate capsules 150mg — Oral dabigatran etexilate mesylate capsules，150mg Once every seven days，two cycle T drug, two cycles R drug

SUMMARY:
In recent years, novel oral anticoagulants (NOACs) such as Factor Xa inhibitors and direct thrombin inhibitors (e.g., dabigatran etexilate) have emerged. These agents target a single factor in the coagulation pathway and offer advantages including rapid onset of action, fixed dosing, no requirement for coagulation monitoring, and fewer interactions with food and other drugs. Their efficacy and safety in patients with non-valvular atrial fibrillation (NVAF) have been validated by large-scale clinical trials.

The aim of this study was to evaluate the bioequivalence of dabigatran mesylate capsules from two different manufacturers after administration to healthy subjects in fasting and postprandial states and to observe the safety of the test and the reference formulation in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects over 18 years old ( including 18 years old ) ;
* Weight index in the range of 19.0 ~ 26.0 kg / m2 ( including the critical value

  * male weight is not less than 50 kg, female weight is not less than 45 kg ;
* Subjects fully understand the purpose, nature, method and possible adverse reactions of the test, volunteer as subjects, and sign informed consent.

Exclusion Criteria:

* The researchers determined that the clinical significance of the cardiovascular system, respiratory system, digestive system, urinary system, endocrine system ;
* Subjects with clinically significant abnormalities in physical examination, vital signs, laboratory tests ( creatinine clearance < 80 mL / min ), 12-lead electrocardiogram ( ECG ), or chest X-ray ( posteroanterior and lateral views ) as deemed by the investigator ;
* Positive results for any of the hepatitis B surface antigen ( HBsAg ), hepatitis B e antigen ( HBeAg ), hepatitis C virus ( HCV ) antibody, human immunodeficiency virus ( HIV ) antibody, or treponema pallidum antibody (TP-Ab) ;
* The investigators determined a history of clinically significant food, drug allergies or other allergic diseases ( asthma, urticaria, eczema dermatitis, etc. ) or any excipients or similar drugs in dabigatran etexilate mesylate capsules have a history of allergy ;
* Subjects with coagulopathy, bleeding tendency ( e.g., recurrent gingival bleeding ), history of bleeding events associated with increased risk within the past 6 months, prior intracranial hemorrhage, gastrointestinal bleeding, purpura, active pathological bleeding, or history of intracranial hemorrhage ;
* Women with a previous history of dysfunctional uterine bleeding, including excessive menstrual bleeding, irregular uterine bleeding, or prolonged menstrual cycles ( length of period > 7 days ) ;
* Patients who underwent surgery within 4 weeks before screening ;
* Those who had a history of drug abuse within 12 months before screening or were positive in urine screening test ;
* Positive alcohol breath test results, or previous alcohol abuse in the past 3 months ( more than 14 units of alcohol per week : 1 unit = beer about 285mL, or spirits about 25mL, or wine about 100mL ), or can not guarantee the test period abandoned drinkers ;
* Patients who drank excessive tea, coffee or caffeine-containing beverages for a long time in the past 3 months ( more than 8 cups a day, 1 cup = 250 mL ), or who drank tea, coffee and / or caffeine-containing beverages within 48 hours before the first administration ;
* Those who have special requirements for diet and cannot comply with a unified diet ( such as intolerance to standard meals, intolerance to lactose, etc. ) or who have difficulty in swallowing, or can not avoid eating grapefruit, grapefruit, mango and other fruits or juices that may affect metabolism ;
* Smokers in the past 3 months ( daily smoking ≥ 5 ) or can not guarantee to give up smoking during the trial ;
* Any prescription drugs, non-prescription drugs, and Chinese herbal medicines were used within 14 days before screening ;
* Anyone who has used any drug that interacts with dabigatran mesylate capsules ( e.g., anticoagulants and antiplatelet aggregating agents, P-gp inhibitors, P-gp inducers, P-gp substrates, other medications affecting P-gp, medications affecting intragastric pH ) in the 4 weeks prior to screening ;
* Those who have participated in a clinical trial of another drug within 3 months prior to screening ( last visit of the previous trial is calculated as the start time ) ;
* Those who have donated ≥ 400mL or 2 units of blood or blood products within 3 months prior to screening or those who have lost ≥ 400mL of blood within 6 months ( except for physiologic blood loss in women ) ;
* Pregnant or breastfeeding women or female subjects who are not using effective contraception within 1 month prior to screening, male subjects ( or their partners ) or female subjects who are planning to become pregnant from the time of signing the informed consent form until 6 months after the last dose, sperm donors or those who are planning to donate eggs, and those who do not wish to use effective contraception during the trial period and for 6 months after the last dose ;
* Those who do not agree to avoid strenuous exercise for 48 hours prior to trial administration ;
* Those who have difficulty in collecting blood intravenously or who suffer from needle and blood sickness ;
* Subjects who, in the opinion of the investigator, are not suitable for participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
maximum observed serum or plasma concentration | 2 day
  The with-subject standard deviation of the pharmacokinetic parameter Cmax of the reference preparation was calculated and the bioequivalence was analyzed according to the bioequivalence evaluation criteria.
area under the serum or plasma concentration-time curve from 0 to t | 2 day
  The with-subject standard deviation of the pharmacokinetic parameter AUC0-t of the reference preparation was calculated and the bioequivalence was analyzed according to the bioequivalence evaluation criteria.
area under the serum or plasma concentration-time curve from 0 to infinity | 2 day
  The with-subject standard deviation of the pharmacokinetic parameter AUC0-inf of the reference preparation was calculated and the bioequivalence was analyzed according to the bioequivalence evaluation criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials Center, The Affiliated Hospital of Guizhou Medical University, Guiyang, China